CLINICAL TRIAL: NCT04671758
Title: Transcatheter Aortic Valve Implantation With Sapien 3 Transcatheter Heart Valve for Pure Aortic Regurgitation. The S3AR Study TAVI With Sapien 3 for Pure AR.
Brief Title: Transcatheter Aortic Valve Implantation With Sapien 3 Transcatheter Heart Valve for Pure Aortic Regurgitation
Acronym: S3AR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI7005J
Record Dates: First submitted 2020-10-15; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-10

CONDITIONS: Pure Aortic Regurgitation
Keywords: pure AR; TAVI; Sapien 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AR TAVI: The population consists in patients with severe symptomatic AR on native aortic valve who are candidates for surgical aortic valve replacement but who are deemed inoperable by the heart team due to technical issues (i.e., porcelain aorta, previous coronary artery bypass grafting,…), extreme left ventricular dysfunction or comorbidities (liver cirrhosis, severe chronic obstructive pulmonary disease…).

SUMMARY:
The hypothesis is that TAVI using a SAPIEN 3 THV is feasible and safe for the treatment of pure AR.

DETAILED DESCRIPTION:
Up to now, the balloon-expandable valves have been considered contraindicated for patients with pure AR due to the absence of calcium which is considered necessary for the anchoring of the prosthesis. Nonetheless, several cases report have suggested the feasibility of TAVI using the SAPIEN XT THV, in patients with no calcified valves suggesting that an appropriate degree of oversizing might compensate the lack of calcium for the anchoring of these prostheses.

The new generation balloon-expandable SAPIEN 3 THV has incorporated changes in the stent frame geometry, leaflets configuration and an external sealing skirt resulting in an increased stability and outstanding control during its implantation, a greater radial force, a reduced rate of paravalvular leaks and a covering of a wider range of annulus dimensions. These characteristics of the SAPIEN 3 THV might translate into a safer use of this device in patients with pure AR and non-calcified valves.

Significant AR occurs in 2.0% of individuals of >75 years, 13.3% of patients referred for intervention, being severe in 5% of these patients. As for aortic stenosis, its prevalence increases with age and the most frequent cause is degenerative although rheumatic and endocarditis are present. Although patients with severe AR have an excess risk of mortality and aortic valve replacement reduces mortality, only 1/3 of patients with significant AR finally undergo intervention. Reasons for no intervention are unknown.

Even if it has been suggested that AR might be underestimated and the prevalence of this disease might be higher than previously reported, and a percent of patients with indication for aortic valve replacement are denied for surgery, pure AR is a small niche of patients for TAVI. In terms of cost-effectiveness, both the development of a dedicated device and the investment in the training of operators in the implantation technique might lack of interest. However, performing TAVI with a device used in the routine practice might be appealing and, importantly, safer. A preliminary case series including 3 patients have suggested the feasibility of TAVI with the SAPIEN 3 device for pure AR (Urena M, Himbert D. JACC, 2016 ). In this study we aim to evaluate the feasibility and long-term safety of the SAPIEN 3 THV in patients with pure AR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic (at least dyspnoea NYHA class III or acute heart failure requiring hospitalisation) and pure AR
* Contraindication or high risk for surgical aortic valve replacement
* Echocardiography and computed tomography findings suitable for TAVI using a SAPIEN 3 THV

Exclusion Criteria:

* Contraindication for TAVI (active endocarditis, aortic dissection, annuloectasia..)
* Patients' refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic (at least dyspnoea NYHA class III or acute heart failure requiring hospitalisation) and pure AR
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and 30-day safety of TAVI with the SAPIEN 3 THV in patients with pure AR | 30 days
  1/ Device success at 1 month follow up according to the Valve Academic Research Consortium (VARC)-2. 2-Rate of moderate or severe AR at 1-month follow-up

SECONDARY OUTCOMES:
Long-term safety of TAVI with the SAPIEN 3 THV in patients with pure AR | 1 year
  Long-term safety defined as lack of valve migration and 1 year cardiovascular mortality defined according to the VARC-2 (combined endpoint)
Long-term performance of TAVI with the SAPIEN 3 THV in patients with pure AR | 1 year
  Rate of moderate or severe AR at 1-year follow-up
Long-term safety of TAVI with the SAPIEN 3 THV in patients with pure AR | 1 year
  Long-term safety defined as lack of 1-year all cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Himbert, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Claude Bernard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Urena M, Himbert D, Ohlmann P, Capretti G, Goublaire C, Kindo M, Morel O, Ghodbane W, Iung B, Vahanian A. Transcatheter Aortic Valve Replacement to Treat Pure Aortic Regurgitation on Noncalcified Native Valves. J Am Coll Cardiol. 2016 Oct 11;68(15):1705-1706. doi: 10.1016/j.jacc.2016.07.746. No abstract available. PMID 27712786